CLINICAL TRIAL: NCT01326195
Title: Dating Violence and HIV Prevention in Girls: Adapting Mental Health Interventions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Christie J. Rizzo Ph.D./Principal Investigator, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K23MH086328 (NIH)
Record Dates: First submitted 2011-03-28; First posted 2011-03-30 (Estimated); Last update posted 2011-03-30 (Estimated); Status verified 2011-03

CONDITIONS: Dating Violence; HIV Infections
Keywords: HIV Prevention; Dating Violence; Females; Romantic relationships; Adolescents; Sexuality; Underserved youth
MeSH Terms: conditions — HIV Infections; Sexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Skills (Experimental): Cognitive-Behavioral Dating Violence and HIV Prevention Group
  Interventions: Behavioral: Cognitive-Behavioral Dating Violence and HIV Prevention Group
- Health Promotion (Active Comparator): Psycho-educational Dating Violence and HIV Prevention group
  Interventions: Behavioral: Psycho-educational Dating Violence and HIV prevention group

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Dating Violence and HIV Prevention Group — Six, two-hour weekly sessions and one 2-hour booster session 6 weeks later with adolescent females
  Other Names: Date SMART
  Arms: Skills
Behavioral: Psycho-educational Dating Violence and HIV prevention group — Knowledge based intervention matched for time and attention to skills arm
  Arms: Health Promotion

SUMMARY:
This project is designed to develop and test a group-based preventive intervention to reduce dating violence and sexual risk behavior among adolescent females with prior dating violence exposure.

DETAILED DESCRIPTION:
A growing body of research reveals that dating violence (DV) plays a significant role in adolescent girls' HIV risk. Dating violence has been associated with less condom use, younger age at first intercourse, having multiple sex partners and alcohol use prior to sexual encounters. Thus, prevention strategies that address dating violence and HIV risk may hold promise for reducing sexual risk behavior among a particularly at-risk population. In this study, a cognitive-behaviorally based intervention named "Skills to Manage Aggression in Relationships for Teens" (Date S.M.A.R.T.) is being developed and compared to a psychoeducational program for dating violence and HIV prevention. The program is being implemented with a sample of underserved youth, as economic disadvantage and minority status have been found to be related to increased rates of adolescent dating violence. A primary focus of the intervention is to address mental health problems (i.e. psychological distress and behavioral dysregulation) that underlie the development and maintenance of both dating violence and sexual risk behavior among adolescent girls.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent must be English-speaking
* Adolescent must have a lifetime history of physical dating violence perpetration or victimization

Exclusion Criteria:

* Current enrollment in an intervention for dating violence or HIV prevention

Ages: 15 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2009-05; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Change in number (#) of unprotected sex acts | Baseline, 3 months, 6 months, 9 months

SECONDARY OUTCOMES:
Change in number of acts of dating violence perpetration and victimization | Baseline, 3 months, 6 months, 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Christie J. Rizzo, Ph.D., Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Rizzo CJ, Joppa M, Barker D, Collibee C, Zlotnick C, Brown LK. Project Date SMART: a Dating Violence (DV) and Sexual Risk Prevention Program for Adolescent Girls with Prior DV Exposure. Prev Sci. 2018 May;19(4):416-426. doi: 10.1007/s11121-018-0871-z. PMID 29352400